CLINICAL TRIAL: NCT03779438
Title: Intramuscular 17-Alpha-Hydroxyprogesterone Caproate for Prevention of Emergent Cesarean Delivery in Symptomatic Pregnant Women With Placenta Previa: A Randomized Controlled Study
Brief Title: 17-Alpha-Hydroxyprogesterone Caproate in Pregnant Women With Placenta Previa
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aswan University Hospital (Other)
Responsible Party: Principal Investigator, hany farouk, Principal Investigator, Aswan University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: aswu/189/18
Record Dates: First submitted 2018-12-15; First posted 2018-12-19 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Placenta Previa
Keywords: cesarean section; placenta previa; antepartum hemorrhage; 17-alpha-Hydroxyprogesterone caproate
MeSH Terms: conditions — Placenta Previa

STUDY DESIGN:
Intervention Model Description: A Double-Blind Randomized Clinical Trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: A Double-Blind Randomized Clinical Trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 17-OHPC (Active Comparator): patients received weekly 250 mg 17 alpha-hydroxyprogesterone-caproate (cidolut depot) intramuscular injections started at 24-26 week and up to 37-weeks' gestation or delivery
  Interventions: Drug: 17-OHPC
- placebo to 17-OHPC (Placebo Comparator): patients received weekly placebo to 17 alpha-hydroxyprogesterone-caproate intramuscular injections started at 24-26 week and up to 37-weeks' gestation or delivery
  Interventions: Drug: placebo to 17-OHPC

INTERVENTIONS:
Drug: 17-OHPC — patients received weekly 250 mg 17 alpha-hydroxyprogesterone-caproate (cidolut depot) intramuscular injections started at 24-26 week and up to 37-weeks' gestation or delivery
  Other Names: Active Comparator; cidolut depot
  Arms: 17-OHPC
Drug: placebo to 17-OHPC — patients received weekly placebo to17 alpha-hydroxyprogesterone-caproate intramuscular injections started at 24-26 week and up to 37-weeks' gestation or delivery
  Other Names: Placebo Comparator
  Arms: placebo to 17-OHPC

SUMMARY:
Purpose to evaluate the effects of intramuscular 17-Alpha-Hydroxyprogesterone Caproate (17-OHPC) for prevention of Emergent Cesarean Delivery in symptomatic Pregnant Women with Placenta Previa

DETAILED DESCRIPTION:
Most authors report an increased risk of bleeding with advancing gestation among women with placenta previa.

The American College of Obstetricians and Gynecologists (ACOG) and the Society for Maternal-Fetal Medicine (SMFM) both recommend the use of 17-OHPC to prevent recurrent spontaneous preterm birth.

Preterm deliveries account for 75% of perinatal mortality and surviving preterm infants are at risk for neurological, respiratory, and gastrointestinal complications. So, it is therefore very important to try to prolong the pregnancy without increasing the risk of emergent delivery in cases with placenta previa. The authors hypothesized that a pharmacological strategy like 17-alpha-Hydroxyprogesterone caproate may improve pregnancy outcomes and may also allow obstetricians to tailor their approach to save delayed scheduled cesarean section women with a placenta previa.

The aim of this study to evaluate the role of17-alpha-Hydroxyprogesterone caproate in the prevention of preterm cesarean delivery (CD) in cases with symptomatic placenta previa with avoids of an emergent CD which affects the maternal outcome and prevents prematurity which affects the prenatal outcome.

ELIGIBILITY:
Inclusion Criteria:

* Estimated gestational age: between 24 weeks and 37 week's gestation
* Confirmed Placenta previa; either major or minor degrees.
* Placenta previa with preterm uterine contractions or with a history of at least single attack of mild vaginal bleeding

Exclusion Criteria:

* Severe attack of bleeding requiring an immediate intervention.
* Fetal heart rates instability or non-reassuring tracing
* Intrauterine fetal death or major fetal anomalies.
* If associated with abruptio placentae
* Patients with known bleeding disorders or on anticoagulant therapy
* Patients with severe medical disorders

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — pregnant women with symptomatic placenta previa
Enrollment: 300 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-03-01 (Estimated)

PRIMARY OUTCOMES:
the duration of prolongation of pregnancy from the time of enrollment to the time of delivery | 6 weeks
  measure the duration of prolongation of pregnancy in days measured from the time of enrollment to the time of delivery

SECONDARY OUTCOMES:
apgar score | 5 minutes postpartum
  measure apgar score from 0 to 10
the number of patients with postpartum hemorrhage | 24 hours post operative
  calculation the number of patients with postpartum hemorrhage

CONTACTS AND LOCATIONS:
Overall Officials: hany f sallam, md, Principal Investigator — Aswan University Hospital
Locations (1):
- Aswan University, Aswān, Egypt

IPD SHARING:
Plan to Share IPD: Undecided